CLINICAL TRIAL: NCT04772820
Title: The SOCIAL Study: Feasibility of Remote Home Support Coaches to Decrease the Physical and Psychological Impact of Social Distancing on Older Adults
Brief Title: Feasibility of Remote Home Support Coaches (SOCIAL Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: University of Maryland, Baltimore (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Shalendar Bhasin, MD, Principal Investigator, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020P004113; 3P30AG031679-10S2 (NIH)
Record Dates: First submitted 2021-02-23; First posted 2021-02-26 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Malnutrition; Isolation; Depression; Anxiety; Sedentary Behavior; Loneliness
Keywords: Covid19; Physical Inactivity; Social Isolation; Inadequate Nutrition; Older Adult; Social Distancing; Remote Home Support; Physical; Psychological; loneliness; behavioral activation
MeSH Terms: conditions — Malnutrition; Depression; Anxiety Disorders; Sedentary Behavior; COVID-19; Social Isolation

STUDY DESIGN:
Intervention Model Description: This project is a single-group unblinded feasibility study to explore a new telephone-based behavioral activation intervention to support homebound older people. If this intervention appears to be feasible, acceptable, and to show preliminary evidence of efficacy the aim will be to evaluate it in a phase III efficacy trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Primary Aim (Other): Brief Behavioral Activation coaching will be delivered by telephone and other remote technology by trained coaches. Over 10 sessions, the coaches will help people to find meaningful activities to decrease loneliness, increase physical activity and improve nutrition.
  Interventions: Behavioral: Telephone-based coaching

INTERVENTIONS:
Behavioral: Telephone-based coaching — A telephone-based brief behavioral activation coaching program that will involve 10 sessions over 4 months. Sessions will focus on helping people to identify meaningful activities that they can safely do to decrease loneliness, increase physical activity and improve nutrition.
  Other Names: Remote coaching

SUMMARY:
The goal of this this study is to develop and test the feasibility of a remotely delivered brief behavioral activation intervention to decrease the negative physical and psychological consequences of being homebound among older adults during the time of COVID.

DETAILED DESCRIPTION:
The goal of this study is to develop and test the feasibility of a remotely delivered brief behavioral activation intervention to decrease the negative physical and psychological consequences of being homebound among older adults during the time of COVID.The intervention will focus on decreasing the impact of social isolation, inactivity and poor nutrition on old people during a time when many in-person social activities are not possible. It will be delivered through telephone and other communication tools that allow remote (i.e. not in person) communication over 10 sessions. Subjects will be a total of 60 people aged 75 years an older, who will be recruited from primary care in the Boston MA region and senior living facilities in the Baltimore MD region. Coaches will be trained using an on-line based modules developed to support this intervention. Self-report outcomes will be measured by telephone at baseline and 4-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* • Men or women who are 75 years or older

  * Must be a patient of Mass General Brigham affiliated with Primary Care Physician departments in Boston, MA OR be a resident of Brightview Senior Living and Assisted Living facilities near Baltimore, MD

Exclusion Criteria:

* • Men or women who are 74 years and younger

  * Participants who are not affiliated with Primary Care Physician departments at Mass General Brigham or a resident of an assisted living facility in Baltimore, MD
  * Unable to adequately complete the Evaluation to Provide Consent

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Physical Activity - Self-report survey to measure engagement in activities | change from baseline to 4-month follow-up
  Yale Physical Activity Survey (self-report)
Loneliness assessment - 20 item, self-report assessment to measure loneliness | change from baseline to 4-month follow-up
  UCLA Loneliness Scale 3.0 (self-report) 20 item, self-report assessment to measure loneliness. Scale from 1(never) to 4(often)
Physical Activity - step activity monitor to track daily steps walked | change in steps from the first week of study to final week (week 16) of study
  average steps walked per day

SECONDARY OUTCOMES:
PROMIS Short form to measure level 2 adult depression | change from baseline to 4-month follow up
  PROMIS Depression (Short Form 8-item, self report)
PROMIS short-form to measure anxiety in adults | change from baseline to 4-month follow up
  PROMIS Anxiety (Short form 8-item, self report)
Late Life Function Instrument to assess functionality in elderly | change from baseline to 4-month follow up
  Late Life Function Instrument (LLFDI - self report)
Late Life Function Instrument to access disability in elderly | change from baseline to 4-month follow up
  Late Life Disability Instrument (LLFDI - self report)
Duke Social Support short scale to measure social support among older people | change from baseline to 4-month follow up
  Duke Social Support Index (self-report)
Mini-nutritional assessment to determine if there is risk of malnourishment | change from baseline to 4-month follow up
  Mini-nutritional assessment - Short Form
Likert 0-7 rating scale of participants satisfaction with the program | 4 month follow-up
  Likert rating of satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Shalender Bhasin, MD, Principal Investigator — Brigham and Women's Hospital; Nancy Latham, PhD, Principal Investigator — Brigham and Women's Hospital; Denise Orwig, PhD, Principal Investigator — University of Maryland, Baltimore
Locations (2):
- United States (2):
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts